CLINICAL TRIAL: NCT01641146
Title: An HIV Intervention for Black Men at Risk
Brief Title: An HIV Intervention for Black Men at Risk - The Enhanced Sexual Health Intervention for Men (ES-HIM)
Acronym: ES-HIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11-000617; 5R34MH077550 (NIH)
Record Dates: First submitted 2012-07-05; First posted 2012-07-16 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: HIV; Depression; Posttraumatic Stress Disorder
Keywords: HIV risk reduction; Stress reduction; Trauma reduction; PTSD
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic | interventions — Menogaril; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Sexual Health Intervention for Men (Experimental): ES-HIM is a six-session intervention for HIV-positive Black bisexual men who have histories of child sexual abuse. Guided by cognitive behavioral approaches and an ecological framework, ES-HIM effects sexual behavior change and psychological health improvement. Sexual risk reduction is framed from the perspective of being a triple minority (i.e., HIV-positive, ethnic and sexual minority). Issues of stigma and social isolation were discussed in regard to these identities. Sexual ownership focusing on individual responsibility for one's health and well-being was prioritized along with caring for sexual partners, family and community. Decisions regarding sexual behaviors and consequences were framed within a culturally congruent social context. Topics included: 1) the influence of gender and ethnicity; (2) early socialization regarding gender and culture, as well as adult experiences; (3) HIV stigma; and (4) recognizing stressors, including histories of personal trauma.
  Interventions: Behavioral: Enhanced Sexual Health Intervention for Men (ES-HIM)
- Health Promotion (HP) Comparison Arm (Active Comparator): Health Promotion Intervention (HP) is the comparison arm. It is designed to control for the Hawthorne effect and reduce the likelihood that effects of ES-HIM could be attributed to special attention and group interaction. HP addresses health issues, including certain cancers, hypertension, diabetes, and heart disease, all of which are common among African American men, but did not focus on sexual behavior. Participants were taught that these diseases could be prevented by changing personal behaviors (e.g., increasing physical activity and healthy dietary practices, ceasing cigarette smoking and alcohol and drug abuse), or managed with early detection and screening behaviors.
  Interventions: Behavioral: Health Promotion (HP) Comparison Arm

INTERVENTIONS:
Behavioral: Enhanced Sexual Health Intervention for Men (ES-HIM) — ES-HIM is a six-session intervention for HIV-positive Black bisexual men who have histories of child sexual abuse. Guided by cognitive behavioral approaches and an ecological framework, ES-HIM effects sexual behavior change and psychological health improvement. Sexual risk reduction is framed from the perspective of being a triple minority (i.e., HIV-positive, ethnic and sexual minority). Issues of stigma and social isolation were discussed in regard to these identities. Sexual ownership focusing on individual responsibility for one's health and well-being was prioritized along with caring for sexual partners, family and community. Decisions regarding sexual behaviors and consequences were framed within a culturally congruent social context. Topics included: 1) the influence of gender and ethnicity; (2) early socialization regarding gender and culture, as well as adult experiences; (3) HIV stigma; and (4) recognizing stressors, including histories of personal trauma.
  Other Names: ES-HIM
  Arms: Enhanced Sexual Health Intervention for Men
Behavioral: Health Promotion (HP) Comparison Arm — Health Promotion Intervention (HP) is the comparison arm. It is designed to control for the Hawthorne effect and reduce the likelihood that effects of ES-HIM could be attributed to special attention and group interaction. HP addresses health issues, including certain cancers, hypertension, diabetes, and heart disease, all of which are common among African American men, but did not focus on sexual behavior. Participants were taught that these diseases could be prevented by changing personal behaviors (e.g., increasing physical activity and healthy dietary practices, ceasing cigarette smoking and alcohol and drug abuse), or managed with early detection and screening behaviors.
  Other Names: HP
  Arms: Health Promotion (HP) Comparison Arm

SUMMARY:
HIV continues to spread among Black men who have sex with men (MSM), but few interventions target high-risk Black men who have sex with men and women (MSMW). Black MSMW with histories of childhood sexual abuse (CSA) may be an especially vulnerable population for: a) high-risk sexual behaviors; b) negative psychological sequelae (e.g., depressive or posttraumatic stress disorder (PTSD) symptoms); and c) neurobiological abnormalities in cardiovascular, neuroendocrine and/or immune systems (e.g., cortisol and norepinephrine), and HIV/AIDS progression. The purpose of this study was to test an HIV risk reduction intervention, guided by the Social Learning Theory, the Ecological Model, and the concept of allostatic load, a composite of the cumulative effects of stress on biological systems including psychoneuroimmunologic markers. The investigators tested the 6-session Enhanced Sexual Health Intervention for Men (ES-HIM) on 88 non-gay identifying HIV-positive Black MSMW with histories of CSA. The outcomes were to reduce high-risk sexual behaviors (i.e., unprotected anal and vaginal sex and number of sex partners) and negative psychological symptoms of depression and PTSD. Links between these outcomes and biomarkers of stress were also explored. Randomization to either the ES-HIM or a health promotion control group occurred with study participants assessed at baseline, post, 3- and 6-months.

DETAILED DESCRIPTION:
The purpose of this small randomized clinical trial was to develop and test the Enhanced Sexual Health Intervention for Men (ES-HIM), designed for non-gay identifying HIV-positive African American MSMW with histories of childhood sexual abuse (CSA). The investigators compared ES-HIM to an attention matched general Health Promotion intervention (HP) on efficacy in reducing: a) sexual risk behaviors (i.e., unprotected anal and vaginal sex and number of sex partners); b) psychological symptoms of PTSD and depression; and c) a biological composite of primary neurohormonal mediators of the stress response (cortisol and catecholamines). The investigators also explored the intervention effects on neopterin, an indicator of HIV disease progression, as an outcome.

Project Aims

1. To determine the impact of the ES-HIM intervention on HIV sexual risk behaviors among non-gay identifying HIV-positive African American men who have sex with men and women (MSMW) who have histories of childhood sexual abuse (CSA). The investigators hypothesize that compared to the Health Promotion comparison condition, the ES-HIM condition will be more effective in decreasing unprotected anal and vaginal sex (i.e., increase condom use) and number of sexual partners at immediate post-intervention and at 3- and 6-months post-intervention.
2. To determine the impact of the ES-HIM intervention on negative psychological symptoms over time among non-gay identifying HIV-positive African American MSMW who have histories of CSA. The investigators hypothesized that compared to the Health Promotion condition, the ES-HIM condition will be more effective in decreasing depressive and posttraumatic stress symptoms at immediate post-intervention and at 3- and 6-months post-intervention.

In addition to these aims, the investigators also explored associations between HIV sexual risk behaviors (i.e., unprotected anal and vaginal sex), negative psychological symptoms (i.e., depressive & posttraumatic stress symptoms) and biomarkers of allostatic load over time among ES-HIM participants.

Research Methods

The University of California, Los Angeles (UCLA) ES-HIM Project was a 4-year study conducted from 2007-2011 to develop and test an HIV risk and stress reduction intervention. Institutional Review Board (IRB) approval for the protection of human subjects in research at UCLA and a Certificate of Confidentiality from the National Institutes of Health (NIH) were obtained.

Intervention Procedures

HIV-positive African American MSMW were recruited through fliers posted at participating community-based organizations, as well as through outreach at community events, bars, clubs, and other locations where the target population may be present. Once interested potential participants were screened and deemed eligible, informed consent was obtained. After informed consent, participants were asked to complete a baseline survey, as well as complete locator forms. Upon completion of the baseline survey, participants were randomized into the ES-HIM active intervention group or the Health Promotion control condition. Both the ES-HIM and the Health Promotion included six sessions, with each session lasting two hours; two sessions were administered per week for three consecutive weeks. The primary aims of the ES-HIM intervention were to increase condom use and decrease symptoms of depression and posttraumatic stress. Within these six, 120-minute sessions, active ES-HIM intervention participants had the opportunity to discuss their sexual experiences and issues of masculinity and stigma associated with being African American, HIV-positive, and a non-gay identifying MSMW. The Health Promotion condition focused on improving general health and concentrated on diet, exercise, relaxation/sleep hygiene, and medication adherence. Both the ES-HIM and Health Promotion curricula were delivered by trained Facilitators.

Data Collection

Enrolled participants were administered surveys via Audio-Computer Assisted Self Interview (A-CASI) at four time points: baseline, immediate post-intervention (upon completion of the sixth ES-HIM or Health Promotion session), and at 3- and 6-months post-intervention. Also, participants were asked to provide 12-hour urine collections for biomarkers of stress and a one time urine sample for neopterin at baseline and 3- and 6-months post-intervention. Non-urinary biomarkers, including height and weight (body mass index), heart rate, blood pressure, and waist-to-hip ratio measurements were collected at these same time points. Data collection (i.e., survey administration, urine container drop-off, and non-urinary biomarker measurements) were administered in confidential settings at collaborative community agencies and/or UCLA.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Male
* English speaking
* HIV-positive
* non-gay identifying
* Black/African American
* Sexually active and engaged in unprotected anal and/or vaginal sex with both a male and female partner in the previous 90 days
* Have a history of child sexual abuse

Exclusion Criteria:

* Younger than 18 years of age
* Female
* Non-English speaking
* HIV-negative or unknown HIV-serostatus
* Race/Ethnicity other than Black / African American
* Not sexually active, uses condoms and/or lacks both male and female partners in past 90 days
* No history of child sexual abuse

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2008-12; Primary Completion 2010-09 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Sexual Risk Behavior Change Over Time - At Three Post Intervention Assessments | Baseline (pre-intervention) and Immediate post, and 3-and 6-months post intervention
  To determine the impact of the ES-HIM intervention on HIV sexual risk behaviors among non-gay identifying HIV-positive African American men who have sex with men and women (MSMW) who have histories of childhood sexual abuse (CSA). The investigators hypothesized that compared to the Health Promotion comparison condition, the ES-HIM condition will be more effective in decreasing unprotected anal and vaginal sex (i.e., increase condom use) and number of sexual partners at immediate post-intervention and at 3- and 6-months post-intervention.
Mental Health Outcome Change Over Time - At Three Post Intervention Assessments | Baseline (pre-intervention) and Immediate post, and 3-and 6-months post intervention
  To determine the impact of the ES-HIM intervention on negative psychological symptoms over time among non-gay identifying HIV-positive African American MSMW who have histories of CSA. The investigators hypothesized that compared to the Health Promotion condition, the ES-HIM condition will be more effective in decreasing depressive and posttraumatic stress disorder symptoms at immediate post-intervention and at 3- and 6-months post-intervention.

SECONDARY OUTCOMES:
Associations between Sexual Risk Behaviors, Mental Health Outcomes and Biomarkers - Changes At Two Post Intervention Assessments | Baseline (pre-intervention) and 3-and 6-month post intervention
  Associations between HIV sexual risk behaviors (i.e., unprotected anal and vaginal sex), negative psychological symptoms (i.e., depressive & posttraumatic stress symptoms) and biomarkers of allostatic load over time among ES-HIM participants will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: John K Williams, MD, Principal Investigator — University of California, Los Angeles
Locations (4):
- United States (4):
  - The AmASSI Health and Cultural Center, Inglewood, California
  - Palms Residential Care Facility, Los Angeles, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - JWCH Institute Inc., Los Angeles, California

REFERENCES:
- [Result] Glover DA, Williams JK, Kisler KA. Using novel methods to examine stress among HIV-positive African American men who have sex with men and women. J Behav Med. 2013 Jun;36(3):283-94. doi: 10.1007/s10865-012-9421-5. Epub 2012 Apr 27. PMID 22538773
- [Result] Williams JK, Glover DA, Wyatt GE, Kisler K, Liu H, Zhang M. A sexual risk and stress reduction intervention designed for HIV-positive bisexual African American men with childhood sexual abuse histories. Am J Public Health. 2013 Aug;103(8):1476-84. doi: 10.2105/AJPH.2012.301121. Epub 2013 Jun 13. PMID 23763412